CLINICAL TRIAL: NCT01251146
Title: Effects of Bisoprolol and Atenolol on Resting Heart Rate and Sympathetic Nervous System's Activity in Patients With Essential Hypertension
Brief Title: A Randomized Controlled Study to Assess the Effects of Bisoprolol and Atenolol on Resting Heart Rate and Sympathetic Nervous System's Activity in Subjects With Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200006-515
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: Hypertension; Bisoprolol; Atenolol
MeSH Terms: conditions — Hypertension | interventions — Bisoprolol; Atenolol

ARMS (2):
- Bisoprolol (Experimental)
  Interventions: Drug: Bisoprolol
- Atenolol (Active Comparator)
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Bisoprolol — Bisoprolol will be administered at a dose of 5 milligram (mg) once daily for 2 weeks. If heart rate is less than or equal to 65 beats per minute (bpm), then the initial dose will be administered for another 2 weeks. If the heart rate remains greater than 65 bpm, then the dose will be further increased to 7.5 mg once daily for 2 weeks. After 2 weeks, if the heart rate is less than or equal to 65 bpm, the increased dose will be administered for another 2 weeks. If the heart rate is still greater than 65 bpm, then the dose will be further increased to 10 mg once daily for 2 weeks. After 2 weeks, if the heart rate is less than or equal to 65 bpm, the increased dose will be administered for another 2 weeks.
  Other Names: Concor®
  Arms: Bisoprolol
Drug: Atenolol — Atenolol will be administered at a dose of 50 mg once daily for 2 weeks. If heart rate is less than or equal to 65 bpm, then the initial dose will be administered for another 2 weeks. If the heart rate remains greater than 65 bpm, then the dose will be further increased to 75 mg once daily for 2 weeks. After 2 weeks, if the heart rate is less than or equal to 65 bpm, the increased dose will be administered for another 2 weeks. If the heart rate still greater than 65 bpm, then the dose will be further increased to 100 mg once daily for 2 weeks. After 2 weeks, If the heart rate is less than or equal to 65 bpm, the increased dose will be administered for another 2 weeks.
  Arms: Atenolol

SUMMARY:
This is a Phase 4, prospective, multi-centric and randomized controlled study to compare the effects of bisoprolol and atenolol on resting heart rate (RHR) and sympathetic nervous system's (SNS) activity in subjects with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 25-65 years
* Subjects with essential hypertension (EH)
* Subjects with systolic blood pressure (SBP) 140-160 millimeter of mercury (mmHg) and diastolic blood pressure (DBP) 90-100 mmHg
* Subjects with normal sinus rhythm
* Subjects with resting heart rate (RHR) greater than 70 bpm
* Subjects who give written informed consent

Exclusion Criteria:

* Subjects with atrial fibrillation (AF)/sick sinus syndrome (SSS)/atrioventricular block II-III Grade (AVB II-III) without pacemaker
* Subjects with bradyarrhythmia/hypotension
* Subjects with unstable angina pectoris (UAP)/acute myocardial infarction (AMI)/heart failure (HF) (New York Heart Association [NYHA] Class III - IV)
* Subjects with uncontrolled diabetes mellitus (DM)
* Subjects with bronchial asthma
* Subjects with gastro-intestinal ulcer or skin ulcer
* Subjects with liver dysfunction/renal impairment
* Subjects treated with calcium channel blockers (except amlodipine) or other beta-blockers.
* Subjects with glaucoma
* Subjects with known allergic/intolerance to beta-blocker
* Pregnant or lactating women
* Subjects who had participated in another clinical study within the last 3 months
* Subjects who have legal incapacity or limited legal capacity

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gao Pingjin, Prof., Principal Investigator — Shanghai Institute of Hypertension
Locations (2):
- China (2):
  - Beijing Shi Jingshan Hospital, Beijing
  - Shanghai Institute of Hypertension, Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- Bisoprolol: Bisoprolol was administered at a dose of 5 milligram (mg) once daily for 2 weeks. If the heart rate was less than or equal to 65 beats per minute (bpm) at Week 2, then the initial dose was administered for another 2 weeks (up to Week 4). If the heart rate was greater than 65 bpm at Week 2, then the dose was further increased to 7.5 mg once daily for 2 weeks (up to Week 4). If the heart rate was less than or equal to 65 bpm at Week 4, the increased dose was administered for another 2 weeks (up to Week 6). If the heart rate was still greater than 65 bpm at Week 4, then the dose was further increased to 10 mg once daily for 2 weeks (up to Week 6). If the heart rate was less than or equal to 65 bpm at Week 6, the increased dose was administered for another 2 weeks (up to Week 8). If the heart rate was still greater than 65 bpm, then the treatment was ceased.
- Atenolol: Atenolol was administered at a dose of 50 mg once daily for 2 weeks. If the heart rate was less than or equal to 65 bpm at Week 2, then the initial dose was administered for another 2 weeks (up to Week 4). If the heart rate was greater than 65 bpm at Week 2, then the dose was further increased to 75 mg once daily for 2 weeks (up to Week 4). If the heart rate was less than or equal to 65 bpm at Week 4, the increased dose was administered for another 2 weeks (up to Week 6). If the heart rate still greater than 65 bpm at Week 4, then the dose was further increased to 100 mg once daily for 2 weeks (up to Week 6). If the heart rate was less than or equal to 65 bpm at Week 6, the increased dose administered for another 2 weeks. If the heart rate was still greater than 65 bpm, then the treatment was ceased.
Period: Overall Study
Arm/Group | Bisoprolol | Atenolol
Started | 86 | 91
Completed | 83 | 81
Not Completed | 3 | 10
Not completed — Lost to Follow-up | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bisoprolol | Atenolol | Total
Number analyzed (Participants) | 86 | 91 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.44 (9.78) | 46.30 (9.87) | 45.88 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 38 | 69
  Male | 55 | 53 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Baroreflex Sensitivity (BRS) at Attainment of Heart Rate Goal
Description: Baroreflex sensitivity (BRS) is an important characteristic of baroreflex control and often noninvasively assessed by relating heart rate (HR) fluctuations to blood pressure (BP) fluctuations. Heart rate goal was defined as attainment of heart rate less than or equal to 65 beats per minute (bpm).
Time Frame: Baseline and attainment of heart rate goal (Week 2 or Week 4 or Week 6)
Population: Intention to treat (ITT) population included all randomized participants who received at least 1 dose of study medication. "N" signifies those participants who were evaluated for this measure. "n" signifies those participants who were evaluated for this measure at the specified time point for each treatment arm group respectively.
Measure: Mean (Standard Deviation); unit: millisecond per millimeter of mercury
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 75 | 79
millisecond per millimeter of mercury
  Baseline (n=75,79) | 7.78 (2.92) | 7.92 (3.26)
  Change at attainment of heart rate goal (n=67,66) | 3.27 (3.67) | 2.88 (4.05)

2. Primary Outcome: Change From Baseline in Baroreflex Sensitivity (BRS) at End of Follow-up
Description: Baroreflex sensitivity (BRS) is an important characteristic of baroreflex control and often noninvasively assessed by relating heart rate (HR) fluctuations to blood pressure (BP) fluctuations. Heart rate goal was defined as attainment of heart rate less than or equal to 65 bpm.
Time Frame: Baseline and end of follow-up (Week 4 or Week 6 or Week 8)
Population: ITT population included all randomized participants who received at least 1 dose of study medication. "N" signifies those participants who were evaluated for this measure.
Measure: Mean (Standard Deviation); unit: millisecond per millimeter of mercury
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 71 | 66
millisecond per millimeter of mercury | 4.08 (3.79) | 3.31 (3.83)

3. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV) for Low Frequency Power (LF) and for High Frequency Power (HF) at Attainment of Heart Rate Goal and End of Follow-up
Description: Heart rate variability (HRV) is used to describe the variations of both instantaneous HR and resting rate (RR) intervals and was evaluated for low frequency power (LF) and for high frequency power (HF). Heart rate goal was defined as attainment of heart rate less than or equal to 65 bpm.
Time Frame: Baseline, attainment of heart rate goal (Week 2 or Week 4 or Week 6) and end of follow-up (Week 4 or Week 6 or Week 8)
Population: ITT population included all randomized participants who received at least 1 dose of study medication. "N" signifies those participants who were evaluated for this measure. "n" signifies those participants who were evaluated for this measure at the specified time point for each treatment arm group respectively.
Measure: Mean (Standard Deviation); unit: millisecond square (ms^2)
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 75 | 79
millisecond square (ms^2)
  HRV for LF at Baseline (n=75,79) | 261.80 (208.40) | 322.09 (315.30)
  Change for LF: heart rate goal (n=71,71) | 90.04 (352.97) | 26.14 (416.51)
  Change at end of follow-up for LF (n=71,66) | 89.40 (330.26) | -22.00 (295.54)
  HRV for HF at Baseline (n=75,79) | 171.26 (161.43) | 193.48 (216.06)
  Change for HF: heart rate goal (n=71,71) | 148.91 (338.13) | 136.67 (314.47)
  Change at end of follow-up for HF (n=71,66) | 186.46 (288.53) | 178.05 (375.70)

4. Secondary Outcome: Change From Baseline in Ratio of Heart Rate Variability (HRV) for Low Frequency Power (LF) to Heart Rate Variability Power (HRV) for High Frequency (HF) (LF/HF) at Attainment of Heart Rate Goal and End of Follow-up
Description: as for outcome 3
Time Frame: Baseline, attainment of heart rate goal (Week 2 or Week 4 or Week 6) and end of follow-up (Week 4 or Week 6 or Week 8)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 75 | 79
ratio
  Baseline (n=75,79) | 2.16 (1.89) | 2.40 (1.96)
  Change at attainment of heart rate goal (n=71,71) | -0.70 (1.76) | -0.90 (1.62)
  Change at end of follow-up (n=71,66) | -0.69 (2.08) | -1.15 (1.68)

5. Secondary Outcome: Number of Participants Attaining Heart Rate Goal at Dosage 1, 2 and 3 of Study Treatment
Description: Dosage 1, 2 and 3 for bisoprolol group was defined as 5 mg, 7.5 mg and 10 mg once daily and for atenolol group as 50 mg, 75 mg and 100 mg once daily, respectively. Heart rate goal was defined as attainment of heart rate less than or equal to 65 bpm.
Time Frame: Baseline up to attainment of heart rate goal (Week 2 or Week 4 or Week 6)
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 86 | 91
participants
  Dosage 1 | 72 | 72
  Dosage 2 | 7 | 6
  Dosage 3 | 1 | 0

6. Secondary Outcome: Percentage of Participants Attaining Heart Rate Goal at Week 2, 4 and 6
Description: Heart rate goal was defined as attainment of heart rate less than or equal to 65 bpm.
Time Frame: Attainment of heart rate goal (Week 2 or Week 4 or Week 6)
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 86 | 91
percentage of participants
  Week 2 | 83.72 [9.41 to 24.81] | 79.12 [13.24 to 29.72]
  Week 4 | 91.86 [3.58 to 15.11] | 85.71 [8.04 to 22.26]
  Week 6 | 93.02 [2.85 to 13.63] | 85.71 [8.04 to 22.26]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: Any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition
Time Frame: Baseline up to end of follow-up (Week 4 or Week 6 or Week 8)
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 86 | 91
participants
  Number of participants with AEs | 6 | 6
  Number of participants with SAEs | 0 | 0

8. Secondary Outcome: Number of Participants Compliant With Study Treatment
Description: Participants compliant with study treatment were the participants who have completed the study treatment regimen.
Time Frame: Baseline up to end of follow-up (Week 4 or Week 6 or Week 8)
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 86 | 91
participants | 83 | 81

ADVERSE EVENTS:
Time Frame: Baseline up to end of follow-up (Week 4 or Week 6 or Week 8)
Arm/Group | Bisoprolol | Atenolol
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/91
Other Adverse Events (participants affected / at risk) | 6/86 | 6/91
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=86) | Atenolol (N=91)
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 1
Elevated Triglyceride (Metabolism and nutrition disorders) | 4 | 4
Elevated Cholesterol (Metabolism and nutrition disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Chest distress (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other